CLINICAL TRIAL: NCT05644015
Title: The Effect of the Education Given With the Escape Room Game on the Learning of Parenteral Drug Administration by Nursing Students.
Brief Title: The Use of Escape Room Game in Nursing Students' Learning About Parenteral Drug Administration.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sakarya University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: Health Sciences
Record Dates: First submitted 2022-11-17; First posted 2022-12-09 (Actual); Last update posted 2022-12-09 (Actual); Status verified 2022-12

CONDITIONS: Gamification
Keywords: Escape room; Gamification; Nursing education

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- experimental group (play group) (Experimental): The experimental group played the escape room game. The experimental group played the game once in total.
  Interventions: Other: escape room game
- control group (No Intervention): No intervention was made in the control group.

INTERVENTIONS:
Other: escape room game — Escape room game is a live action team based game where players discover clues, solve puzzles and complete tasks in one or more rooms to accomplish a specific goal (usually by escaping the room) in limited time.
  Arms: experimental group (play group)

SUMMARY:
This study was conducted as a randomized controlled experimental design with a pretest-posttest control group in order to determine the effect of the education given to nursing students with the escape room game on the students' learning of parenteral drug administration. 72 students enrolled in Nursing Fundamentals II Course in the Spring Semester of 2021-2022 Academic Year at Gazi University Faculty of Health Sciences Nursing Department were included in this study. The students were divided into two groups, 36 control and 36 experimental, by randomization method. Written permission was obtained from the ethics committee and the institution in order to conduct the study. Data were collected with "Descriptive Characteristics Form", "Parenteral drug administration Knowledge Test", "Parenteral drug administration Checklists" and "Game Evaluation Form". The first knowledge (pre-test) and skills (Objective structured clinical exam=OSCE) were measured after the parenteral drug administration theoretical course and the skill course in the laboratory were given to the sample group. The sample group was assigned to the experimental and control groups according to the first knowledge and skill measurements. The experimental group played the escape room game in groups of 4 each. The control group was given the right to work independently in the laboratory. The game was played once in the experimental group. Then, the final knowledge (post-test) and final skills (OSCE) of the experimental and control groups were measured. Independent sample t test, chi-square test, Pearson correlation test and dependent sample t test were used to evaluate the data.

DETAILED DESCRIPTION:
First of all, after the theoretical course of parenteral drug administration was explained to the students in the control and experimental groups by the researchers, the course was applied on model patients in the skill laboratory of the faculty. Then, the knowledge and skills of both the experimental and control groups were measured. The knowledge of the students was measured by the knowledge test prepared by the researchers. The skills of the students were evaluated with the OSCE exam by using a checklist by instructors other than the researchers. Afterwards, the 'escape room' game was played by the researchers in the skill laboratory of the faculty with the experimental group. The control group, on the other hand, was given the right to work independently in the faculty's skill laboratory to perform the skills related to the subject. After the game, the knowledge and skills of both the experimental and control groups were measured again. The knowledge of the students was measured by the knowledge test prepared by the researchers. The skills of the students were evaluated with the OSCE exam by using a checklist by instructors other than the researchers. The game was played once with the experimental group. For the game, the experimental group (36) was divided into 9 groups of 4 people each. In the game, each student was expected to perform the related skill of the patient (model patient) in the related patient room in the skill laboratory, and to perform the activities (puzzle, puzzle, etc.) in the patient rooms together as a group.

Escape room game is a type of social game that requires groups of four to ten people to work together based on solving a series of puzzles to escape from a locked room. Although the escape room game is a social game, it has been used in education and training in the last few years. The game features puzzles that students must solve in a limited time to open the box by placing a set of locks on a closed box. Participants work together to find and solve clues around the room to unlock each of the locks.

Preparation of the escape room:

Gazi University Faculty of Health Sciences nursing basics skills laboratory has been transformed into an escape room. In order for the first year students to gain knowledge and skills about parenteral drug applications and reach their learning goals, four patient rooms in which parenteral drug administration skills are practiced in clinical order were created in the skill laboratory and made ready for the escape room game. In order for students to perform activities and skills related to the subject; locked chest box, number coded chest lock, stopwatch, blackboard, whistle, materials to be used in puzzle making, colored paper and cardboard, etc., on which activity questions are processed. Along with the materials, the medical materials (injector, sharps-drilling waste box, cotton, gloves, etc.) that the students will use while performing their parenteral drug administration skills were provided by the researchers.

In each patient room, model patient, patient bed, arm-hip model, bedside unit, bedside table, bedside table; nurse file and related activities developed by the researchers were placed. Curtains and screens were used to separate each patient bed from each other in order to create a patient room layout. The treatment car, which will be used to prepare the treatment of the patients, was placed in an area suitable for the skill laboratory by placing the necessary materials inside. In addition, a locked box and a whiteboard were placed in a suitable area in the middle of the skills lab. In this way, a clinical environment was created and the escape room was made ready. Escape room game rules were created by the researchers in order to determine the game limits and for the participants to understand the game easily.

ELIGIBILITY:
Inclusion Criteria:

* Enrolling for the first time in Nursing Fundamentals II Course,
* Being willing to participate in the research

Exclusion Criteria:

* Having a high school, associate or undergraduate degree in a health-related field,
* It is the inability to use the Turkish language effectively.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2022-05-25 (Actual); Primary Completion 2022-05-28 (Actual); Study Completion 2022-06-15 (Actual)

PRIMARY OUTCOMES:
Measuring the knowledge level of the sample group | two days before randomization
  The knowledge levels of all students participating in the study were measured with the 'parenteral drug administration knowledge test'.
  The students (n:72) participating in the study were randomly assigned to the experimental (n:36) and control (n:36) groups according to their knowledge levels.
Measuring the skill levels of the sample group | two days before randomization
  The skill levels of all students participating in the study were measured with 'parenteral drug administration checklists'.

SECONDARY OUTCOMES:
measuring the knowledge levels of the experimental and control groups | two weeks after starting the intervention (post escape room game)
  After playing the escape room game, the knowledge level of the experimental group was measured with the 'parenteral drug administration knowledge test'.
  The knowledge level of the control group was measured with the 'parenteral drug administration knowledge test'.
measuring the skills of the experimental and control groups | two weeks after starting the intervention (post escape room game)
  skills of the experimental group after playing the escape room game measured with the 'parenteral drug administration checklist'. The skills of the control group were measured with the 'parenteral drug administration checklist'.

CONTACTS AND LOCATIONS:
Overall Officials: Nurhan Aktaş, Principal Investigator — researcher
Locations (1):
- Gazi University, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Darby W, Bergeron P, Brown N, DeFoor M, Jones B. Escape Room Relay Race: "Go for the Gold" in Formative Assessment. J Nurs Educ. 2020 Nov 1;59(11):646-650. doi: 10.3928/01484834-20201020-09. PMID 33119778
- [Result] Roman P, Rodriguez-Arrastia M, Molina-Torres G, Marquez-Hernandez VV, Gutierrez-Puertas L, Ropero-Padilla C. The escape room as evaluation method: A qualitative study of nursing students' experiences. Med Teach. 2020 Apr;42(4):403-410. doi: 10.1080/0142159X.2019.1687865. Epub 2019 Nov 18. PMID 31738615